CLINICAL TRIAL: NCT06409637
Title: A Prospective, Single-arm Clinical Study of FOLFOX Combined With Lenvatinib as Adjuvant Chemotherapy to Prevent Tumor Recurrence After Liver Transplantation for Hepatocellular Carcinoma Beyond Milan Criteria
Brief Title: FOLFOX Plus Lenvatinib Adjuvant Therapy for Hepatocellular Carcinoma Post-Liver Transplantation
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SYSKY-2024-167-01
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Liver Cancer; Liver Transplant
MeSH Terms: conditions — Liver Neoplasms | interventions — Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOX plus Lenvatinib (Experimental): FOLFOX4 regimen: Oxaliplatin 85mg/m2 intravenous infusion over 2 hours on Day 1; Leucovorin 400mg/m2 intravenous infusion over 2 hours on Days 1-2; 5-Fluorouracil (5-FU) initially 400mg/m2 intravenous bolus followed by 2400mg/m2 continuous intravenous infusion over 46 hours. Each cycle lasts for 4 weeks, repeated every 4 weeks for a total of 6-8 cycles.
  Lenvatinib: For patients with a body weight <60 kg, the recommended daily dose of lenvatinib is 8 mg (2 capsules of 4 mg each), once daily; for patients with a body weight ≥60 kg, the recommended daily dose of lenvatinib is 12 mg (3 capsules of 4 mg each), once daily. Treatment should be continued until disease progression, intolerable adverse effects, or the end of the study.
  Interventions: Drug: FOLFOX4 regimen; Drug: lenvatinib

INTERVENTIONS:
Drug: FOLFOX4 regimen — FOLFOX4 regimen: Oxaliplatin 85mg/m2 intravenous infusion over 2 hours on Day 1; Leucovorin 400mg/m2 intravenous infusion over 2 hours on Days 1-2; 5-Fluorouracil (5-FU) initially 400mg/m2 intravenous bolus followed by 2400mg/m2 continuous intravenous infusion over 46 hours. Each cycle lasts for 4 weeks, repeated every 4 weeks for a total of 6-8 cycles.
  Other Names: Oxaliplatin, Leucovorin, 5-Fluorouracil
Drug: lenvatinib — Lenvatinib: For patients with a body weight <60 kg, the recommended daily dose of lenvatinib is 8 mg (2 capsules of 4 mg each), once daily; for patients with a body weight ≥60 kg, the recommended daily dose of lenvatinib is 12 mg (3 capsules of 4 mg each), once daily. Treatment should be continued until disease progression, intolerable adverse effects, or the end of the study.
  Other Names: lenvatinib pill

SUMMARY:
Liver transplantation not only removes the liver tumor (seed) but also eliminates the underlying diseased liver (soil), making it an essential therapeutic approach for hepatocellular carcinoma (HCC). However, the tumor recurrence post-liver transplantation significantly jeopardizing the long-term survival of transplant recipients. Given the scarcity of donor livers, exploring effective measures to prevent tumor recurrence after liver transplantation holds significant clinical and societal value. Currently, there is no consensus on adjuvant therapy for preventing tumor recurrence post-liver transplantation for HCC, and the quantity and quality of studies on systemic chemotherapy are limited. In recent years, administration of the FOLFOX regimen combined with lenvatinib has been widely used in the treatment of advanced HCC, showing remarkable efficacy. The aim of this study is to investigate the efficacy and safety of adjuvant chemotherapy with FOLFOX combined with lenvatinib in preventing tumor recurrence after liver transplantation for HCC beyond Milan criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years inclusive.
2. Histologically confirmed hepatocellular carcinoma without other non-hepatocellular carcinoma components.
3. ECOG performance status 0-1.
4. Child-Pugh class A liver function.
5. Eligible for chemotherapy and targeted therapy within 1-2 months after liver transplantation.
6. Immunosuppressive regimen including calcineurin inhibitors, mycophenolate mofetil, and sirolimus.
7. Adequate liver, kidney, and bone marrow function: serum albumin >28g/L, total bilirubin ≤3mg/dL (51.3 umol/l), ALT and AST ≤5 times the upper limit of normal; serum creatinine ≤1.5 times the upper limit of normal; hemoglobin >90g/L, absolute neutrophil count (ANC) >1.5×10^9/L, platelet count >60×10^9/L; PT-INR <1.5 or PT within normal limits +6 seconds.
8. Negative serum/urine pregnancy test within 7 days prior to treatment initiation for fertile women.
9. Reliable contraception must be used by all male and female participants during the trial and for six months after its completion.
10. Ability to take oral medications.
11. Participants must provide written informed consent.

Exclusion Criteria:

1. Life expectancy less than 6 months.
2. High suspicion of hepatocellular carcinoma recurrence and metastasis.
3. Concurrent malignancies.
4. Allergy to lenvatinib or chemotherapy drugs.
5. Pregnant or lactating women (female participants must undergo pregnancy testing within 7 days prior to treatment).
6. History of severe cardiovascular diseases: congestive heart failure >NYHA class 2; active coronary artery disease (myocardial infarction within 6 months prior to enrollment); severe arrhythmias requiring antiarrhythmic therapy (β-blockers or digoxin permitted); uncontrolled hypertension.
7. History of HIV infection.
8. Severe active clinical infections.
9. Patients requiring medication for epilepsy (e.g., steroids or antiepileptic drugs).
10. Patients with kidney diseases requiring dialysis.
11. Drug abuse, medical conditions, psychiatric illnesses, or social status that may interfere with the participant's participation in the study or evaluation of study results.
12. Patients unable to swallow oral medications, such as those with severe upper gastrointestinal obstruction requiring gastric tube feeding.
13. Previous treatment with other anti-angiogenic therapies, surgery, TACE, local therapy, systemic chemotherapy, immunotherapy, etc., before liver transplantation.
14. Clear evidence of main portal vein/hepatic vein tumor thrombus or inferior vena cava tumor thrombus.
15. Clear evidence of lymph node metastasis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 62 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival | 2 years
  From the date of transplantation to the date of tumor recurrence or the date of tumor progression otherwise, with censoring at the date of death or last contact for event-free patients.

SECONDARY OUTCOMES:
2-year overall survival | 2 years
  The cumulative incidence of patients surviving the next 2 years from the start of treatment.
Adverse event and validation of adverse event incidence | 2 years
  The grade and incidence of adverse events (including laboratory tests, vital signs, electrocardiogram and other safety-related indicators, especially hematological system toxicity, liver transplantation function impairment, etc.) during the study, as well as the incidence of serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Leibo Xu, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Organ Transplantation Center, Sun Yat-sen Memorial Hospital, Sun Yat-sen University,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No